CLINICAL TRIAL: NCT01840267
Title: The Effect of Pneumoperitoneum on Intracranial Pressure in Pediatric Laparoscopic Surgery: Ultrasonographic Measurement of Optic Nerve Sheath Diameter
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0090
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Intracranial Pressure
Keywords: pneumoperitoneum; pediatric laparoscopy; optic nerve sheath diameter; intracranial pressure
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- laparoscopic surgery under general anesthesia: pediatric patients undergoing laparoscopic surgery under general anesthesia
  Interventions: Device: ultrasonographic measurement of optic nerve sheath diameter

INTERVENTIONS:
Device: ultrasonographic measurement of optic nerve sheath diameter — A thick layer of gel is applied on the upper closed eyelid. The linear 13- to 6-MHz ultrasound probe is then placed in the gel, without exerting pressure on the eye. Two measurements are taken for each optic nerve: one in the transverse plane, with the probe being horizontal, and one in the sagittal plane, with the probe being vertical. The final ONSD is the mean of these measurements.

SUMMARY:
The pneumoperitoneum during laparoscopic surgery in pediatrics has the potential to cause an increase of intracranial pressure (ICP). Previous studies have proposed that ultrasonographic measurements of the optic nerve sheath diameter (ONSD) correlate with signs of increased ICP. Therefore, this study aims to confirm the increased ICP by ultrasonographic measurement of ONSD during laparoscopic surgery in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. pediatric patients (under 9 yrs) scheduled for undergoing laparoscopic surgery under general anesthesia

Exclusion Criteria:

1. Patients with previous history of neurologic disease or neurosurgery, ocular disease or ocular surgery

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients undergoing laparoscopic surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
ultrasonographic measurement of optic nerve sheath diameter | change of ultrasonographic measurement of optic nerve sheath in 10 minutes after anesthesia induction, 10 minutes after pneumoperitoneum, and 10 minutes after CO2 desufflation.
  A thick layer of gel is applied on the upper closed eyelid. The linear 13- to 6-MHz ultrasound probe is then placed in the gel, without exerting pressure on the eye. Two measurements are taken for each optic nerve: one in the transverse plane, with the probe being horizontal, and one in the sagittal plane, with the probe being vertical. The final ONSD is the mean of these measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Seoul, Seoul, South Korea